CLINICAL TRIAL: NCT00923169
Title: A Phase 1 Study of the Safety and Efficacy of GC1008: A Human Anti-Transforming Growth Factor-Beta (TGFBeta) Monoclonal Antibody in Patients With Advanced Renal Cell Carcinoma or Malignant Melanoma
Brief Title: Part 2 of Phase 1 Study of GC1008 to Treat Advanced Melanoma (Part 2 Will Only Accept and Treat Patients With Advanced Malignant Melanoma)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060200; 06-C-0200; NCT00899444 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2012-06-29

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell; Melanoma; Monoclonal Antibodies; Phase I; TGF-B
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma

INTERVENTIONS:
Drug: Anti-Transforming Growth Factor-beta (GC 1008)

SUMMARY:
Background:

* GC1008 is a genetically engineered antibody designed to block the activity of transforming growth factor-beta (TGF-beta). Although TGF-beta has some normal and beneficial effects in the body, it is often over-produced in malignant melanoma tumors, and it can help the melanoma grow and spread.
* Part 1 of this study enrolled 22 subjects with malignant melanoma or kidney cancer to determine the highest safe dose of GC1008, which was found to be 15 mg/kg.
* Three of 22 patients with malignant melanoma in Part 1 of the study developed skin problems, but it is not known if these problems were related to the administration of GC1008.

Objectives:

-To determine the frequency of adverse skin side effects of GC1008 in patients with malignant melanoma.

Eligibility:

-Patients 18 years of age and older with malignant melanoma for whom previous treatment was not successful.

Design:

* GC1008 is given intravenously (through a vein) at a dose of 15 mg/kg or 10 mg/kg for four doses on study days 0, 28, 42 and 56 (one treatment cycle). Patients whose cancer responds to GC1008 may receive one or two additional treatment cycles of four doses given every two weeks.
* Physical exam and vital signs on study days 1, 14, 28, 42, 56, 84 and 140.
* Vitals signs on study days 0, 14, 28, 42, 56, 84 and 140.
* Frequent blood sample collections for routine safety tests, measurement of blood levels of GC1008, analysis for antibodies against GC1008 and for research studies.
* CT or MRI scan, bone scan and PET CT scan before treatment and on study day 84 and 140.
* Biopsy of apparently normal skin before treatment and again on day 84.
* Review of medicines and well being on study days 0, 14, 28, 42, 56, 84, 112 and 140.
* Follow-up visits every 3 months for up 2 years for patients who have not received additional treatment for their cancer. Evaluations include physical exam, CT or MRI scan, PET CT scan, blood tests and possibly tumor biopsies.

DETAILED DESCRIPTION:
BACKGROUND:

Transforming growth factor-beta (TGFBeta) is a member of a large family of evolutionarily conserved proteins with broad activity.

Paradoxically, TGFBeta is involved in both preventing malignant transformation of cells and promoting tumor progression by enhancing the proteolysis of extracellular matrix, stimulating tumor cell migration, tumor invasiveness, angiogenesis and inhibiting the immune response to tumor.

GC1008 is a human IgG4 monoclonal antibody that neutralizes all isoforms of TGFBeta.

GC1008 reduced metastatic burden and enhanced immune responses against cancers in preclinical studies.

OBJECTIVES:

To assess the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and safety of GC1008 in patients with locally advanced of metastatic renal cell carcinoma or malignant melanoma.

To obtain pharmacokinetic (PK) and pharmacodynamic data on GC1008.

To evaluate tumor response as a preliminary assessment of clinical activity.

To assess possible surrogate markers that might predict clinical efficacy by obtaining tumors and blood samples for exploratory biomarker analysis.

ELIGIBILITY:

Adult patients with locally advanced, surgically inoperable metastatic renal cell carcinoma or malignant melanoma. The Part 2 cohort expansion will accrue only malignant melanoma patients.

Patients must have failed greater than or equal to 1 prior therapy.

Patients must have a hemoglobin greater than or equal to 10.0 gm/dL granulocyte count (ANC) of greater than or equal to 1500/miocroliter and platelets greater than or equal to 100,000/microliter; creatinine less than or equal to 2 mg/dL, serum bilirubin less than or equal to 1.5 x ULN, meet criteria for AST/ALT and have a normal PT/PTT.

Measurable disease by RECIST criteria.

Patients must test negative for hepatitis B virus, hepatitis C virus and human immune deficiency virus (HIV).

Patient must be greater than 4-weeks since major surgery, radiation therapy or chemotherapy.

DESIGN:

Part 1: Cohorts of 3-6 patients will be treated with a single intravenous dose of GC1008 at doses of 0.1 to 15 mg/kg as prescribed by the protocol (This part has been completed).

Part 2: A cohort expansion will treat an additional 6 subjects with GC1008 15 mg/kg to estimate the frequency of unacceptable skin adverse events (e.g., keratoacanthomas, etc). If an unacceptable frequency of skin adverse events are observed, an additional 6 subjects will be treated at the lower dose of 10 mg/kg to determine the phase II dose.

Patients will then be observed for adverse events and PK studies obtained for 4-weeks.

Patients will then receive three additional doses of GC1008 at same dose every 2-weeks. Responding patients and those with stable disease may receive additional treatments.

ELIGIBILITY:
* All inclusion and exclusion criteria must be met and confirmed prior to enrollment. Unless specified, all laboratory normal ranges that are mentioned in inclusion and exclusion criteria refer to institutional criteria. Unless otherwise specified, all inclusion, exclusion and patients withdrawal criteria apply to both Part 1 and Part 2 of this Phase 1 study.

INCLUSION CRITERIA:<TAB>

1. In Part 1, Dose Escalation: Patients with histologically confirmed, locally advanced and surgically inoperable or metastatic renal cell carcinoma or malignant melanoma are eligible.

   In Part 2, Patient Expansion: Patients with histologically confirmed, locally advanced and surgically inoperable or metastatic malignant melanoma are eligible.

   In both Parts 1 and 2: All patients must have failed greater than or equal to 1 prior therapy and potential patients may not be eligible for curative intent treatment (e.g., potentially curative surgical resection or chemotherapy). Other qualifying therapies include any medical, surgical, radiation, or investigational approach used for potential therapeutic benefit (but not for diagnostic purposes) in patients with advanced disease.

   In addition, in Part 1, patients with renal cell carcinoma must have failed temsirolimus and either sorafenib or sunitinib as part of their prior therapies.
2. Age greater than or equal to 18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2.
4. Serum albumin greater than or equal to 3.0 g/dL.
5. Expected survival greater than or equal to 5 months.
6. Adequate organ function including:

   1. Marrow: Hemoglobin greater than or equal to 10.0 g/dL, absolute neutrophil count (ANC) greater than or equal to 1,500/mm(3), and platelets greater than or equal to 100,000/mm(3).
   2. Hepatic: Serum total bilirubin less than or equal to 1.5 x upper limit of normal (ULN) (Patients with Gilberts's Disease may be included if their total bilirubin is less than or equal to 3.0 mg/dL), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 2.5 x ULN. If the patient has known liver metastases, an ALT and/or AST less than or equal to 5 x ULN are allowed.
   3. Renal: If negative proteinuria on urine dipstick, serum creatinine (sCR) less than 2 mg/dL or urine creatinine clearance greater than or equal to 60 mL/min. If urine is 1+ positive (30 mg/dL), urine protein must be less than or equal to 1 g/24 hours and measured creatinine clearance greater than or equal to 60 mL/min.
   4. Other: Prothrombin time (PT) and partial thromboplastin time (PTT) within normal ranges.
7. Measurable disease. Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) within 4 weeks prior to first dose of GC1008 (tumor lesion must be new or progressive if in a previously irradiated region.
8. Patients must have negative test (antibody and /or antigen) for hepatitis viruses B and C and human immunodeficiency virus (HIV), unless the result is consistent with prior vaccination or prior infection with full recovery.
9. At the time of enrollment, patients must be greater than 4 weeks since major surgery, radiotherapy, chemotherapy (greater than or equal to 6 weeks if they were treated with a nitrosourea, mitomycin, or monoclonal antibodies such as bevacizumab), immunotherapy, or biotherapy/targeted therapies and recovered from the toxicity of prior treatment to less than or equal to Grade 1, exclusive of alopecia. Concurrent cancer therapy is not permitted. (In patients who received long-acting agents, a treatment-free interval of 2 half-lives should be considered.)
10. Patients must be able to give written informed consent to participate. Patients may not be consented by a durable power of attorney.
11. Male and female patients of child-producing potential must agree to use effective contraception while enrolled on study and receiving the experimental drug, and for at least 3 months after the last treatment. Female patients of child-producing potential must have a negative serum pregnancy test confirmed within 7 days of receiving the initial dose of GC1008 therapy.
12. Documentation of flu vaccination if enrolled during flu season (as defined by the availability of vaccine). Otherwise, patients should receive the current flu vaccine greater than or equal to 1 week before beginning GC1008 therapy.
13. Pre-treatment tumor samples, such as paraffin blocks or unstained slides, must be available for analyses.

EXCLUSION CRITERIA:

1. Central nervous system (CNS) metastases, meningeal carcinomatosis, malignant seizures, or a disease that either causes or threatens neurologic compromise (e.g., unstable vertebral metastases).
2. History of ascites or pleural effusions, unless successfully treated, completely resolved, and the patient has not been treated for these conditions for greater than 4 months.
3. Active thrombophlebitis, thromboembolism, hypercoagulability states, bleeding, or use of anti-coagulation therapy (including anti-platelet agents). Patients with a history of deep venous thrombosis may participate if successfully treated, completely resolved, and no treatment has been given for greater than 4 months.
4. Hypercalcemia: Calcium greater than 11.0 mg/dL (2.75 mmol/L) unresponsive or uncontrolled in response to standard therapy (e.g., bisphosphonates).
5. Pregnant or nursing women, due to the unknown effects of GC1008 on the developing fetus or newborn infant.
6. Patients diagnosed with another malignancy - unless following curative intent therapy, the patient has been disease free for at least 5 years and the probability of recurrence of the prior malignancy is less than 5 percent. Patients with curatively treated early-stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia (CIN) are eligible for this study.
7. Patients with an organ transplant, including those that have received an allogeneic bone marrow transplant.
8. Use of investigational agents within 4 weeks prior to study enrollment (within 6 weeks if the treatment was with a long-acting agent such as a monoclonal antibody).
9. Patients on immunosuppressive therapy including:

   1. Systemic corticosteroid therapy for any reason, including replacement therapy for hypoadrenalism. Patients receiving inhaled or topical corticosteroids may participate.
   2. Patients receiving cyclosporine A, tacrolimus, or sirolimus are not eligible for this study.
10. Significant or uncontrolled medical illness, such as congestive heart failure (CHF), myocardial infarction, symptomatic coronary artery disease, significant ventricular arrhythmias within the last 6 months, or significant pulmonary dysfunction. Patients with a remote history of asthma or active mild asthma may participate.
11. Active infection, including unexplained fever (temperature greater than 38.1 YC), or antibiotic therapy within 1 week prior to enrollment.
12. Systemic autoimmune disease (e.g., systemic lupus erythematosus, active rheumatoid arthritis, etc.).
13. A known allergy to any component of GC1008.
14. Patients who, in the opinion of the Investigator, have significant medical or psychosocial problems that warrant exclusion. Examples of significant problems include, but are not limited to:

    1. Other serious non-malignancy-associated medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis) or significantly increase the risk of SAEs.
    2. Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up, or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment.).
    3. Patients currently abusing drugs or alcohol or, in the opinion of the Investigator, at high for poor compliance.
15. Part 2 only: Prior therapy with a TGFBeta antagonist, such as an antibody, receptor, or kinase inhibitor or anti-sense therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-07-09; Primary Completion 2010-01-20 (Actual); Study Completion 2010-01-20 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and safety of GC1008 in patients with locally advanced or metastatic renal cell carcinoma or malignant melanoma.

SECONDARY OUTCOMES:
To obtain pharmacokinetic (PK) and pharmacodynamic (PD) data on GC1008.

CONTACTS AND LOCATIONS:
Overall Officials: Jay A Berzofsky, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Cancer Institute of New Jersey, Little Brunswick, New Jersey, United States

REFERENCES:
- [Background] Bandyopadhyay A, Zhu Y, Cibull ML, Bao L, Chen C, Sun L. A soluble transforming growth factor beta type III receptor suppresses tumorigenicity and metastasis of human breast cancer MDA-MB-231 cells. Cancer Res. 1999 Oct 1;59(19):5041-6. PMID 10519421
- [Background] Blobe GC, Schiemann WP, Lodish HF. Role of transforming growth factor beta in human disease. N Engl J Med. 2000 May 4;342(18):1350-8. doi: 10.1056/NEJM200005043421807. No abstract available. PMID 10793168
- [Background] Derynck R, Akhurst RJ, Balmain A. TGF-beta signaling in tumor suppression and cancer progression. Nat Genet. 2001 Oct;29(2):117-29. doi: 10.1038/ng1001-117. PMID 11586292